CLINICAL TRIAL: NCT01608321
Title: rTMS for the Treatment of Chronic Pain in GW1 Veterans
Acronym: rTMS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Did not meet recruitment goals
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPLD-001-11F
Record Dates: First submitted 2012-05-25; First posted 2012-05-31 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; Gulf War Illness; Gulf War Syndrome; Fibromyalgia; repetitive Transcranial Magnetic Stimulation; Transcranial Magnetic Stimulation; Veterans
MeSH Terms: conditions — Chronic Pain; Persian Gulf Syndrome; Fibromyalgia

STUDY DESIGN:
Intervention Model Description: Double-blind study of rTMS versus sham
Who Masked: Participant, Care Provider, Investigator
Masking Description: rTMS sham involves using the same paddle applied to the head, the side (one shielded internally from the magnetic pulse by aluminum) turned toward the head is randomized. A small shock is also given in both circumstances to disguise the sensation produced by the active rTMS.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rTMS (Experimental): Those receiving experimental treatment will receive 20 sessions of rTMS. The treatment will be delivered by trained medical personnel.
  Interventions: Device: rTMS
- Sham rTMS (Placebo Comparator): Those receiving the sham rTMS will receive 20 sessions of sham rTMS. The treatment will be delivered by trained medical personnel.
  Interventions: Device: Sham device

INTERVENTIONS:
Device: rTMS — Repetitive Transcranial Magnetic Stimulation
  Arms: rTMS
Device: Sham device — Placebo Device that simulates active rTMS treatment
  Arms: Sham rTMS

SUMMARY:
This study was designed to evaluate the effect of repetitive Transcranial Magnetic Stimulation (rTMS) in the resolution of Chronic Pain. Participants will be Veterans from the first Gulf War (GW1) who often suffer from chronic pain problems.

DETAILED DESCRIPTION:
A number of studies have been conducted on the health of Veterans deployed to Iraq during GW1. The focus of these studies has been primarily to define the nature of symptoms and symptom clusters and to determine if evidence supports the definition of a new unique illness. Most noteworthy is the "Iowa Study", a cross-sectional study of 3,695 Veterans from Iowa consisting of those who were and were not deployed in GW1. In telephone interviews the Gulf War deployed Veterans reported approximately twice the number of symptoms compared to those who were not deployed.

The often ambiguous and seemingly treatment resistant symptoms presented by GW1 Veterans represent a challenge to the Veteran's Affairs Health Care System on two fronts; efficacy in treatment and cost. In particular, unlike most medical conditions which can be diagnosed by objective medical findings, pain is a subjective experience (International Association for the Study of Pain, 1994). Therefore the investigators propose to engage in a clinical trial of rTMS in chronic pain that occurs in the context of multiple medical symptoms in the GW1 population. The symptom category approach will be applied with the restriction that enrolled GWI diagnosed patients will have symptoms of chronic pain as outlined in the musculoskeletal category and at least two additional symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Born between 1936 and 1973 (ages 18 to 55 during Gulf War I) and were deployed to the Persian Gulf during Gulf War I.
* Patients must have symptoms suggestive of Gulf War Illness, including

  * Chronic pain >= 4 on the pain severity scale of the BPI-SF at screening
  * At least 2 other symptoms in at least one of the other five (5) categories defined by the 2013 IOM report (Gulf War and Health, Treatment for Chronic Multisymptom Illness): fatigue, mood and cognition, gastrointestinal, respiratory, and neurological
* Ability to obtain a Motor Threshold (MT) will be determined at the end of the screening process.
* If on a psychotropic medication regimen, that regimen will be stable for at least 4 weeks prior to entry to the study and patient will be willing to remain on a stable regimen during the acute treatment phase.
* Has an adequately stable condition and environment to enable attendance at scheduled clinic visits.
* For female participants, agrees to use one of the following acceptable methods of birth control:

  * Complete abstinence (not having sexual intercourse with anyone)
  * An oral contraceptive (birth control pills)
  * Norplant
  * Depo-Provera
  * A condom with spermicide
  * A cervical cap with spermicide
  * A diaphragm with spermicide
  * An Intrauterine device
  * Surgical sterilization (having your tubes tied)
* Able to read, verbalize understanding and voluntarily sign the Informed Consent Form prior to performance of any study-specific procedures or assessments.

Exclusion Criteria:

* Pregnant or lactating female (This is a Federal Drug Administration (FDA)-required exclusion. In the future, if rTMS becomes a proven treatment for pain, its safety in the context of pregnancy should be studied separately (Nahas et al 1999)).
* Unable to be safely withdrawn, at least two-weeks prior to treatment commencement, from medications that substantially increases the risk of having seizures.
* Have a cardiac pacemaker.
* Have an implanted device (deep brain stimulation) or metal in the brain.
* Have a mass lesion, cerebral infarct or other active central nervous system (CNS) disease, including a seizure disorder.
* Known current psychosis as determined by Diagnostic and Statistical Manual (DSM-IV) coding in chart (Axis I, psychotic disorder, schizophrenia) or a history of a non-mood psychotic disorder.
* Diagnosis of Bipolar Affective Disorder (as determined by chart review and intake interview)
* Current amnesic disorders, dementia, Mini Mental Status Exam (MMSE) 24 or delirium.
* Current substance abuse (not including caffeine or nicotine) as determined by positive toxicology screen, or by medical history, within 3 months prior to screening.
* History of loss of consciousness greater than 15 minutes due to head injury.
* Participation in another concurrent clinical trial.
* Patients with prior exposure to rTMS.
* Active current suicidal intent or plan. Patient at risk for suicide will be required to establish a written safety plan involving their primary psychiatrist and the treatment team before entering the clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-09; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W Ashford, MD PhD, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
Trial discontinued before an adequate number of subjects was tested.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | rTMS | Sham rTMS
Started | 13 | 4
Completed | 12 | 4
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rTMS | Sham rTMS | Total
Number analyzed (Participants) | 13 | 4 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 4 | 17
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 10 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 10 | 4 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 10 | 3 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in the Brief Pain Inventory (Short Form) Score
Description: The Brief Pain Inventory (BPI) is one of the most widely used measurement tools for assessing clinical pain. The BPI allows patients to rate the severity of their pain and the degree to which their pain interferes with common dimensions of feeling and function. The basic pain scale rating is a rating of 0-10 with 0 as no pain, and 10 the worst pain imaginable.
Time Frame: Comparison of baseline BPI and end-of-treatment BPI (time 3-4 weeks)
Population: One patient did not meet study entry criteria at baseline (pain scale score = 0), so was not included in the analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | rTMS | Sham rTMS
Number analyzed (Participants) | 11 | 4
units on a scale | -1.2 (1.5) | -.9 (1.6)

ADVERSE EVENTS:
Arm/Group | rTMS | Sham rTMS
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/4
Other Adverse Events (participants affected / at risk) | 2/13 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rTMS (N=13) | Sham rTMS (N=4)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Elevated blood glucose = 600, considered unrelated to treatment.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rTMS (N=13) | Sham rTMS (N=4)
headache (General disorders) | 1 (6) | 0 (0) — post-rTMS headache
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — blood sugar = 153 (known diabetic)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No